CLINICAL TRIAL: NCT04692688
Title: Randomized, Placebo-Controlled, Double-Masked Study of the Safety and Efficacy of Orally Administered APX3330 in Subjects With Moderately Severe to Severe Non-Proliferative Diabetic Retinopathy and Mild Proliferative Diabetic Retinopathy
Brief Title: Study of the Safety and Efficacy of APX3330 in Diabetic Retinopathy
Acronym: ZETA-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocuphire Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPI-APXDR-201 (ZETA-1)
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema; NPDR - Non Proliferative Diabetic Retinopathy; PDR - Proliferative Diabetic Retinopathy
Keywords: diabetes; diabetic retinopathy; NPDR; PDR
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This is a placebo-controlled, double-masked, randomized, Phase 2 study in approximately 100 subjects with moderately severe to severe non-proliferative diabetic retinopathy (NPDR), or mild proliferative diabetic retinopathy (PDR), evaluating safety and efficacy following administration of APX3330 twice daily for 24 weeks.
  The study will have a 1:1 randomization (placebo: APX3330). Randomization will be stratified by level of disease severity (NPDR or PDR). Subjects with mild PDR will be capped at 20% for each arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- APX3330 (Experimental): Five 120 mg tablets will be taken by mouth as follows: 3 tablets every morning and 2 tablets every evening.
  Interventions: Drug: APX3330
- Placebo (Placebo Comparator): Five 120 mg tablets will be taken by mouth as follows: 3 tablets every morning and 2 tablets every evening.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APX3330 — APX3330, a small-molecule oral tablet, is a Ref-1 inhibitor that can potentially reduce proinflammatory and hypoxic signaling that contributes to several eye diseases.
  Arms: APX3330
Drug: Placebo — Placebo tablets are identical to APX3330 tablets except for the absence of the active pharmaceutical ingredient.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of APX3330 to treat diabetic retinopathy (DR) and diabetic macular edema (DME).

DETAILED DESCRIPTION:
The objective of this study is to evaluate the efficacy of APX3330 to improve Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Score (DRSS) in one hundred (100) subjects with moderately severe to severe NPDR or mild PDR.

Subjects with moderately severe to severe NPDR and mild PDR will be selected for study participation and be screened for study eligibility.

The eligible eye with the highest DRSS, as assessed by the central reading center, will be designated as the study eye for the primary efficacy analysis.

If the subject meets all eligibility criteria, then the subject will be randomized into the study and receive study medication. Blood will be drawn for biomarker analysis.

The total length of subject participation is approximately 26 weeks, with 5 clinic visits, 4 telephone safety calls, and one telephone call follow-up visit.

The execution of the entire study (first subject screen through last randomized subject completed) is expected to be approximately 12 to 15 months.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant females ≥ 18 years of age
2. At least one eye with DR graded at least moderately severe to severe NPDR or mild PDR (corresponding to DRSS 47, 53, or 61)
3. BCVA assessed by ETDRS protocol letters score of ≥ 60 letters (Snellen equivalent ≥ 20/63)
4. Body mass index (BMI) between 18 and 40 kg/m2, inclusive

Exclusion Criteria:

Ophthalmic:

1. Any prior treatment in the study eye with:

   1. Focal or grid laser photocoagulation within the past year or PRP at any time
   2. Systemic or intravitreal anti-VEGF agents within the last 6 months
   3. Intraocular steroids including triamcinolone and dexamethasone implant within the last 6 months
   4. Fluocinolone implant within the last 3 years
2. Active uveitis, vitritis, or infection in either eye including infectious conjunctivitis, keratitis, scleritis, or endophthalmitis.
3. Ocular incisional surgery including cataract surgery in the study eye within 3 months.
4. Clinically significant ocular disease in either eye.
5. Presence of macular or retinal vascular disease including diabetic macular edema, retinopathy from causes other than diabetes, age-related macular degeneration, pattern dystrophy, choroidal neovascularization of any cause, retinal vein occlusion, retinal artery occlusion in the study eye.
6. History of retinal detachment, full-thickness macular hole in the study eye, or idiopathic or autoimmune uveitis in either eye.

Systemic:

1. Known hypersensitivity or contraindication to study drug.
2. Any disease or medical condition that in the opinion of the Investigator would interfere with the study, prevent the subject from successfully participating in the study, or which might confound the study results.
3. Participation in any investigational study within 30 days prior to screening or planning to participate in any other investigational drug or device clinical trials within 30 days of study completion.
4. Resting HR outside the specified range (50-110 beats per minute).
5. Known to be immunocompromised or receiving immunosuppressive therapy.
6. Hypertension with resting diastolic blood pressure (BP) > 105 mmHg or systolic BP > 200 mmHg.
7. History of chronic liver disease or presence of elevated alanine aminotransferase (ALT) and aspartate aminotransferase (AST) consistent with such diagnosis.
8. Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Percent of Subjects with an improvement in Diabetic Retinopathy Severity Score (DRSS) | 24 Weeks
  Percent of subjects with a ≥ 2-step improvement in DRSS in the study eye

SECONDARY OUTCOMES:
Percent of Subjects with change in Diabetic Retinopathy Severity Scale (DRSS) Scores | Up to 24 Weeks
  Percent of subjects with an improvement or worsening in DRSS of ≥ 1, ≥ 2, ≥ 3, and ≥ 4 steps at Week 12 and Week 24
Mean Change in Diabetic Retinopathy Severity Scale (DRSS) Score | 24 Weeks
  Mean change from baseline in DRSS at Week 24. DRSS is scored on a range from 10 to 90 with 13 discrete scores given within that range and where higher scores indicate a worse outcome.
Percent of Subjects without DR/DME Disease Progression | 24 Weeks
  Percent of subjects not developing center-involved DME or moderate PDR or PDR-related AEs during the study at Week 12 and Week 24
Mean Change in Best-Corrected Visual Acuity (BCVA) | 24 Weeks
  Mean change in BCVA at Week 24
Mean Change in Central Subfield Thickness (CST) | 24 Weeks
  Mean Change in CST at Week 24

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Clinical Site 9, Phoenix, Arizona
  - Clinical Site 8, Bakersfield, California
  - Clinical Site 5, Beverly Hills, California
  - Clinical Site 11, Palm Desert, California
  - Clinical Site 2, Sacramento, California
  - Clinical Site 24, Walnut Creek, California
  - Clinical Site 19, Miami, Florida
  - Clinical Site 7, Winter Haven, Florida
  - Clinical Site 6, Carmel, Indiana
  - Clinical Site 14, Hagerstown, Maryland
  - Clinical Site 22, Springfield, Massachusetts
  - Clinical Site 17, Grand Blanc, Michigan
  - Clinical Site 12, Albuquerque, New Mexico
  - Clinical Site 15, Shirley, New York
  - Clinical Site 20, Charlotte, North Carolina
  - Clinical Site 1, Rapid City, South Dakota
  - Clinical Site 18, Austin, Texas
  - Clinical Site 16, Bellaire, Texas
  - Clinical Site 10, Fort Worth, Texas
  - Clinical Site 4, McAllen, Texas
  - Clinical Site 3, San Antonio, Texas
  - Clinical Site 23, San Antonio, Texas
  - Clinical Site 13, Southlake, Texas
  - Clinical Site 21, Ogden, Utah